CLINICAL TRIAL: NCT05699668
Title: Preterm Infants REtinalMicrovascular Alterations by Means of OCT Angiography
Acronym: PREMA-OCTA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PREMA-OCTA
Record Dates: First submitted 2022-12-14; First posted 2023-01-26 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2022-07

CONDITIONS: Premature With Dysplasia Bronchopulmonary; Premature Without Dysplasia Bronchopulmonary; Controls Born at Term

STUDY DESIGN:
Intervention Model Description: Premature infants born at a term ≤28 weeks of amenorrhea, without bronchopulmonary dysplasia (BPD), whether or not followed at CHIC Premature infants born at a term ≤28 weeks of amenorrhea, with bronchopulmonary dysplasia (BPD) and followed or not at CHIC Patients in the control group (without prematurity without BPD) selected at a scheduled routine ophthalmology consultation at CHIC, born at a term ≥ 38SA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- older premature children born at a term ≤28 weeks of amenorrhea without dysplasia bronchopulmonary (Experimental): OCT Angiography
  Interventions: Device: OCT Angiography
- older premature children born at a term ≤28 weeks of amenorrhea with dysplasia bronchopulmonary (Experimental): OCT Angiography
  Interventions: Device: OCT Angiography
- patients in the control group without prematurity without BPD (Experimental): OCT Angiography
  Interventions: Device: OCT Angiography

INTERVENTIONS:
Device: OCT Angiography — 2 views per eye (one centered on the fovea, one centered on the optic nerve), in 6x6 mm, using the OCT-A Plexelite®.
  Acquisition time per image: about 10 seconds.

SUMMARY:
Retinal vascularization in humans develops between the 16th and 36th week of amenorrhea, centrifugally from the papilla. In case of premature birth, the immature retinal periphery is at risk of ischemic damage due to lack of vascular development.

Prematurity is often associated with respiratory fragility. It often requires ventilatory assistance in the form of oxygen therapy, invasive (oro-tracheal intubation) or non-invasive, which leads to reflex arteriolar vasoconstriction aggravating the ischemia already present. One may wonder if there are subclinical retinal vascular changes, detectable on Tomographie par Cohérence Optique-Angiography (, that could explain the greater risk of amblyopia and optical correction observed. Tomographie par Cohérence Optique-Angiography is a fast growing technique in retinal vascular pathologies: it is a simple, fast, reliable, non-invasive, injection-free examination, which allows to study in high resolution the retinal vascularization, with a distinct analysis of the retinal plexuses and the choriocapillaris

DETAILED DESCRIPTION:
Retinal vascularization in humans develops between the 16th and 36th week of amenorrhea, centrifugally from the papilla. In case of premature birth, the immature retinal periphery is at risk of ischemia due to lack of vascular development. This lack of perfusion in the retinal periphery leads to abnormal secretion of pro-angiogenic factors, promoting the appearance of abnormal neovessels, which can be complicated by intravitreal hemorrhage and tractional retinal detachment, permanently altering vision.

Conversely, it is known that in premature infants, there is a smaller central avascular zone compared to full-term infants. This area of the retina, where 90% of the cones are concentrated, must be free of vascular structures to allow optimal vision.

Prematurity is often associated with respiratory fragility. It often requires ventilatory support in the form of oxygen therapy, invasive (oro-tracheal intubation) or non-invasive, which causes reflex arteriolar vasoconstriction, aggravating the ischemia already present in the periphery.

Clinically, after birth, ocular disorders are more frequently found in preterm infants: amblyopia and contrast vision disorders, ametropia, strabismus and optic nerve anomalies.

It is questionable whether there are subclinical retinal vascular changes, detectable on Tomographie par Cohérence Optique-Angiography, associated with clinical differences.

Indeed, Angiography-Tomographie par Cohérence Optique allows detection of changes in foveolar and peripapillary retinal microvascularization more sensitively than dilated fundus examination (detection of subclinical microvascular abnormalities), as has been demonstrated for many retinal pathologies; it thus participates in the diagnosis, monitoring, evaluation of therapeutic response and prognosis of many retinal Angiography Tomographie par Cohérence Optique is rapidly expanding in retinal vascular pathologies: it is a simple, rapid, reliable, noninvasive, and injection-free examination that allows high-resolution study of the retinal vasculature, with a distinct analysis of the retinal plexuses and the choriocapillaris.

It would also be interesting to investigate whether there is a correlation between the child's neonatal parameters, the retinal vascular changes on Angiography -Tomographie par Cohérence Optique, and the elements of the clinical examination (vision and refraction). If such a correlation is found, it would allow a targeted and personalized visual screening of the subjects identified as most at risk, with a stratification of the ocular risk according to the neonatal history and the OCT-A measurements.

Finally, this study would provide a better understanding of the development of the retina during the neonatal period, the factors that may influence it, and the mechanisms potentially responsible for the observed disorders.

ELIGIBILITY:
Inclusion Criteria:

Premature group:

- Any child aged 5 to 15 years born before or at 28 SA (with or without BPD), followed or not at the Creteil's hospital intercommunal

Control group:

* Any child aged 5 to 15 years born ≥ 38SA, consulting ophthalmology at the Creteil 's hospital intercommunal.
* Acceptance to participate in the protocol
* Child living near the Creteil's intercommunal hospital
* Affiliated to a social security system

Exclusion Criteria: all groups

* Neurobehavioral disorder or psychomotor delay that does not allow the examination to be performed
* Presence of a POR with zone I involvement or having received IVT of anti-VEGF (as it may directly modify the OCT-A parameters)
* Pre-existing retinal pathology: macular scarring of any etiology, retinal vascular alterations such as sickle cell disease, diabetes.
* Pre-existing optic nerve pathologies: glaucoma, coloboma, tumors.
* Chronic respiratory pathologies other than BPD (i.e. not associated with prematurity): cystic fibrosis, DDB...
* General pathology unrelated to prematurity that may have a retinal impact: e.g. respiratory diseases other than BPD
* Participation in an interventional study in ophthalmology
* A history of hyperthermic convulsions in infants or epilepsy, which contraindicates the use of eye drops.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
To show a difference on vascular density in OCT-A (%), between preterm children (born ≤ 28 SA) and control children (born > 38SA). | 1day
  Macular and peripapillary vascular densities (%):on OCT-A images at the superficial and deep capillary plexus in the control and preterm groups

SECONDARY OUTCOMES:
To demonstrate differences in clinical parameters (visual acuity, spherical equivalent) between premature children (born ≤ 28 SA) and control children (born > 38SA) | 1 day
  Collection of clinical parameters
To demonstrate differences in OCT-A parameters (fractal dimension), between premature children (born ≤ 28 SA) and control children (born > 38SA) | 1 day
  Collection of clinical parameters
To demonstrate a correlation between neonatal history (term, birth weight, duration of oxygen therapy, ventilation mode, presence or absence of BPD), clinical parameters (visual acuity, spherical equivalent), and OCT-A parameters. | 1 day
  Collection of neonatal history
To demonstrate differences in OCT-A parameters (central avascular zone area (mm2), between premature children (born ≤ 28 SA) and control children (born > 38SA) | 1 day
  Collection of OCT angiography parameters

IPD SHARING:
Plan to Share IPD: No